CLINICAL TRIAL: NCT01710787
Title: A Phase III, Multi-Center, Randomized, Double-Blind, Parallel-Groups Clinical Trial Comparing the Efficacy and Safety of Intranasally Administered Kovacaine Mist to Tetracaine Alone and to Placebo for Anesthetizing Maxillary Teeth in Adults
Brief Title: Comparison of Intranasal Kovacaine Mist, Tetracaine Alone, and Placebo for Anesthetizing Maxillary Teeth in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Triligent International (Industry); Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SR 3-02
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia
Keywords: operative; dental procedure
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kovacaine Mist, 3 sprays unilateral (Experimental): Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
- Tetracaine Only, 3 sprays unilateral (Experimental): Tetracaine HCl 3%
  Interventions: Drug: Tetracaine HCl 3%
- Placebo, 3 sprays unilateral (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% — 3 unilateral intranasal sprays per dose
  Other Names: Kovacaine Mist
  Arms: Kovacaine Mist, 3 sprays unilateral
Drug: Tetracaine HCl 3% — 3 unilateral intranasal sprays per dose
  Other Names: Active control
  Arms: Tetracaine Only, 3 sprays unilateral
Drug: Placebo — 3 unilateral intranasal sprays per dose
  Other Names: Inactive ingredients
  Arms: Placebo, 3 sprays unilateral

SUMMARY:
The purpose of this study is to compare the efficacy of Kovacaine Mist, Tetracaine only, and Placebo for inducing pulpal anesthesia of the maxillary teeth in adults.

DETAILED DESCRIPTION:
The study will employ a multi-center, randomized, double-blind, placebo-controlled, parallel-groups design to assess the safety and efficacy of Kovacaine Mist delivered intranasally for inducing pulpal anesthesia of maxillary teeth numbers 4 to 13 (maxillary right second premolar to maxillary left second premolar) sufficient to allow completion of the Study Dental Procedure.

The intent is to treat 110 subjects, with enrollment balanced evenly between the 2 study sites, 2:2:1 randomization within each study site and an overall goal of 44 subjects treated with Kovacaine Mist, 44 treated with Tetracaine alone, and 22 treated with Placebo. Recruitment will be from diverse dental patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older.
* Need for an operative restorative dental procedure requiring local anesthesia for a single vital maxillary tooth (other than a maxillary first, second, or third molar) with no evidence of pulpal pathology.
* Normal lip, nose, eyelid, and cheek sensation.
* Able to understand and sign the study informed consent document, communicate with the investigators, and understand and comply with the requirements of the protocol.
* Patency of the naris ipsilateral to the tooth undergoing the Study Dental Procedure.
* Resting heart rate (HR) between 55 and 100 beats per minute (bpm), inclusive.
* Seated systolic blood pressure (SBP) between 95 and 140 mm Hg, inclusive and seated diastolic blood pressure (DBP) between 60 and 90 mm Hg, inclusive.

Exclusion Criteria:

* Inadequately controlled hypertension (blood pressure greater than 140/90 mm Hg).
* Inadequately controlled active thyroid disease of any type.
* Frequent nose bleeds (≥ 5 per month).
* Having received dental care requiring a local anesthetic within the last 24 hours.
* History of allergy to or intolerance of tetracaine, benzyl alcohol, other ester local anesthetics, or para-aminobenzoic acid (as found in PABA-containing sunscreen).
* History of allergy or hypersensitivity to articaine, oxymetazoline, epinephrine, or sulfite preservatives.
* Use of a monoamine oxidase inhibitor within the 3 weeks preceding study entry.
* Nursing, pregnant, suspected of being pregnant, or trying to become pregnant. (Females of child-bearing potential will be required to take a urine pregnancy test on the day of, but prior to, study drug administration to rule out pregnancy.)
* Having received any investigational drug and/or participation in any clinical trial within 30 days prior to study participation.
* Having used oxymetazoline or phenylephrine nasal spray, nasal irrigation, or other nasal or oral decongestant on the day of the study procedure.
* History of congenital or idiopathic methemoglobinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Moore, DMD/PhD/MPH, Study Director — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Buffalo, Buffalo, New York
  - Family and Cosmetic Dentistry, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ciancio SG, Marberger AD, Ayoub F, Garlapo DA, Pantera EA Jr, Pantera CT, Al-Mubarak S, Sobieraj BD, He DY, Myneni SR. Comparison of 3 intranasal mists for anesthetizing maxillary teeth in adults: A randomized, double-masked, multicenter phase 3 clinical trial. J Am Dent Assoc. 2016 May;147(5):339-347.e1. doi: 10.1016/j.adaj.2015.11.009. Epub 2016 Feb 15. PMID 26892312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Started | 44 | 44 | 22
Completed | 44 | 44 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral | Total
Number analyzed (Participants) | 44 | 44 | 22 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (14.73) | 31.3 (12.01) | 35.7 (14.64) | 34.5 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 16 | 12 | 58
  Male | 14 | 28 | 10 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Study Dental Procedure After Without Need for Rescue by Injection of Local Anesthetic.
Description: If the participant does not have sufficient anesthesia to complete the Study Dental Procedure, the participant is given a rescue injection of local anesthetic and is considered a failure for this outcome.
Time Frame: at 15 minutes with a 3 minute window
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
percentage of patients | 84.1 [69.9 to 93.4] | 27.3 [15 to 42.8] | 27.3 [10.7 to 50.2]

2. Secondary Outcome: Intraoral Soft-tissue Anesthesia (Yes/no)
Description: Number of patients who reported no pain when incisive papilla soft-tissue was tested with a probe at designated timepoints
Time Frame: at Baseline, 15, 30, 45, 60, 90, and 120 minutes with a 3 minute window
Population: Only patients from one site (out of the two sites for the study) are used for this analysis. The other site administered this assessment incorrectly.
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 24 | 24 | 12
Participants
  Baseline | 0 | 0 | 0
  15 mins | 19 | 8 | 0
  30 mins | 17 | 3 | 0
  45 mins | 21 | 5 | 3
  60 mins | 17 | 2 | 1
  90 mins | 10 | 1 | 0
  120 mins | 5 | 0 | 0

3. Secondary Outcome: Number of Participants With a Heart Rate Higher Than 125 Bpm
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
Participants | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With a Heart Rate Lower Than 50 Bpm
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
Participants | 1 | 2 | 0

5. Secondary Outcome: Number of Participants With an Increase From Baseline in Systolic Blood Pressure Greater Than or Equal to 25 mm Hg and to a Value Higher Than 160 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
Participants | 2 | 1 | 0

6. Secondary Outcome: Number of Participants With a Decrease From Baseline in Systolic Blood Pressure Greater Than or Equal to 15 mm Hg and to a Value Lower Than 90 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With an Increase From Baseline in Diastolic Blood Pressure Greater Than or Equal to 15 mm Hg and to a Value Higher Than 105 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
Participants | 1 | 0 | 0

8. Secondary Outcome: Number of Participants With a Decrease From Baseline in Diastolic Blood Pressure Greater Than or Equal to 10 mm Hg and to a Value Lower Than 50 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
participants | 1 | 0 | 0

9. Secondary Outcome: Absolute Maximum Change From Baseline in Heart Rate
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
bpm | 9.4 (11.53) | 10.5 (10.74) | 7.0 (7.97)

10. Secondary Outcome: Absolute Maximum Change From Baseline in Systolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
mm Hg | 13.7 (10.74) | 10.8 (9.15) | 5.1 (9.32)

11. Secondary Outcome: Absolute Maximum Change From Baseline in Diastolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
mmHg | 10.5 (7.12) | 7.3 (4.96) | 6.7 (4.91)

12. Secondary Outcome: The Profile Over Time of Heart Rate
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
beats per minute
  Pre-Study (Baseline) | 76.5 (13.10) | 75.1 (10.25) | 74.8 (10.65)
  10 mins | 75.3 (19.25) | 76 (12.03) | 76.3 (12.88)
  30 mins | 69.8 (17.52) | 82.6 (10.81) | 76.0 (17.15)
  45 mins | 72.8 (16.76) | 74.1 (9.40) | 73.1 (12.35)
  60 mins | 71.3 (17.81) | 73.2 (12.03) | 73.0 (10.95)
  90 mins | 73.1 (18.79) | 72.0 (13.12) | 72.1 (11.44)
  120 mins | 71.4 (15.51) | 73.8 (12.37) | 73.7 (9.92)

13. Secondary Outcome: The Profile Over Time of Systolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
mmHg
  Pre-Study (Baseline) | 121.3 (12.09) | 118.6 (10.15) | 118.5 (11.76)
  10 mins | 125.0 (12.49) | 122.0 (13.01) | 121.5 (14.44)
  30 mins | 123.5 (16.65) | 122.2 (14.06) | 130.5 (5.45)
  45 mins | 121.7 (14.2) | 125.1 (12.12) | 118.7 (14.17)
  60 mins | 123.1 (14.16) | 121.7 (13.14) | 117.5 (11.40)
  90 mins | 124.3 (15.55) | 122.1 (16.30) | 116.6 (10.76)
  120 mins | 125.0 (15.75) | 121.1 (12.97) | 115.7 (9.36)

14. Secondary Outcome: The Profile Over Time of Diastolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
mmHg
  Pre-Study (Baseline) | 75.0 (7.92) | 75.3 (8.25) | 74.8 (7.20)
  10 mins | 79.6 (10.44) | 77.7 (8.36) | 77.3 (9.29)
  30 mins | 81.7 (10.91) | 79.6 (10.16) | 84.5 (5.51)
  45 mins | 77.1 (9.06) | 78.7 (9.03) | 75.4 (9.73)
  60 mins | 79.0 (10.63) | 76.8 (9.01) | 76.6 (7.33)
  90 mins | 79.3 (10.91) | 75.7 (8.56) | 74.1 (5.42)
  120 mins | 77.8 (8.85) | 76.9 (8.84) | 75.7 (6.83)

15. Secondary Outcome: Alcohol Sniff Test
Description: The distance from the nose (in centimeters) that a patient is able to detect the smell of alcohol on an alcohol swab.
Time Frame: administered at baseline, 120 minutes and approximately 24 hours after drug administration
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 44 | 44 | 22
cm
  Pre-Study (Baseline) | 19.2 (8.96) | 18.8 (10) | 21.2 (8.35)
  120 Minutes | 18 (9.47) | 17.7 (9.48) | 20.9 (8.13)
  24 Hours | 18.2 (8.51) | 16.1 (8.74) | 20.4 (8.38)

16. Secondary Outcome: Intraoral Soft-tissue Anesthesia (Onset and Duration)
Description: Mean onset and duration of incisive papilla anesthesia based on number of patients who reported no pain when soft-tissue was tested with a probe at designated timepoints
Time Frame: up to 120 mins post-dose
Population: The analysis population includes patients who received a rescue injection of local anesthetic. Local anesthetic may cause soft-tissue anesthesia, impacting this endpoint. In addition, only patients from one site (out of the two sites for the study) are used for this analysis. The other site administered this assessment incorrectly.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 24 | 24 | 12
minutes
  Onset | 9.7 (7.5) | 19.5 (17.6) | 37.0 (0.0)
  Duration | 79.2 (27.0) | 32.1 (15.2) | 26.0 (17.3)

ADVERSE EVENTS:
Time Frame: 24 hours post-dosing
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/44 | 0/22
Other Adverse Events (participants affected / at risk) | 42/44 | 44/44 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kovacaine Mist, 3 Sprays Unilateral (N=44) | Tetracaine Only, 3 Sprays Unilateral (N=44) | Placebo, 3 Sprays Unilateral (N=22)
Cellulitis Orbital (Infections and infestations) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kovacaine Mist, 3 Sprays Unilateral (N=44) | Tetracaine Only, 3 Sprays Unilateral (N=44) | Placebo, 3 Sprays Unilateral (N=22)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 16 | 0 — (runny nose)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 27 | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 1
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 0 — (throat numbness)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Headache (Nervous system disorders) | 6 | 1 | 1
Lacrimation increased (Eye disorders) | 7 | 4 | 0 — (tearing or watery eyes)
Hypertension (Vascular disorders) | 4 | 1 | 1
Intranasal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 2
Toothache (Gastrointestinal disorders) | 2 | 10 | 5 — (Dental Pain, usually attributed to insufficient anesthesia)
Bradycardia (Cardiac disorders) | 4 | 2 | 1
Tachycardia (Cardiac disorders) | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No